CLINICAL TRIAL: NCT06607965
Title: Effects of Whey Protein Combined With Carbohydrates in the ERAS Protocol on the Recovery of Thyroid Cancer Patients After Lateral Neck Dissection: A Prospective Cohort Study
Brief Title: Whey Protein and Carbohydrates in ERAS for Recovery After Thyroidectomy: A Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY S2023-039-01
Record Dates: First submitted 2024-09-13; First posted 2024-09-23 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Whey Protein; Thyroid Neoplasms; Neck Dislocation; Enhanced Recovery After Surgery
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Whey Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Experimental Group:
  6 hours before surgery, patients orally consumed 250 ml of a full-nutrition liquid (220 ml homogenized diet, 50 g; containing 31.4 g carbohydrates, 8 g protein, and 215 kcal).
  2 hours before surgery, patients orally consumed 200 ml of a clear liquid (50 g enzymatically hydrolyzed rice powder + 0.5 g low-sodium salt; containing 47.7 g carbohydrates, 6.5 g whey protein, and 193 kcal).
  After surgery, once there were no symptoms such as dizziness or vomiting, patients could start consuming clear liquids (containing 47.7 g carbohydrates, 6.5 g protein, and 221 kcal) orally every 30 minutes, 4 times on the day of surgery.
  Starting from the first day after surgery, patients consumed 200 ml of fat-free nutritional liquid (50 g enzymatically hydrolyzed rice powder + 7.5 g isolated whey protein + 0.5 g low-sodium salt; 223 kcal) per serving, 4 to 6 times per day as needed.
  Interventions: Dietary Supplement: Whey Protein and Carbohydrates
- control group (No Intervention): Patients fasted for 12 hours before surgery, and after surgery, intravenous fluids were administered. Fat-free diet began after 24 hours post-surgery.

INTERVENTIONS:
Dietary Supplement: Whey Protein and Carbohydrates — Experimental Group:
  6 hours before surgery, patients orally consumed 250 ml of a full-nutrition liquid (220 ml homogenized diet, 50 g; containing 31.4 g carbohydrates, 8 g protein, and 215 kcal).
  2 hours before surgery, patients orally consumed 200 ml of a clear liquid (50 g enzymatically hydrolyzed rice powder + 0.5 g low-sodium salt; containing 47.7 g carbohydrates, 6.5 g whey protein, and 193 kcal).
  After surgery, once there were no symptoms such as dizziness or vomiting, patients could start consuming clear liquids (containing 47.7 g carbohydrates, 6.5 g protein, and 221 kcal) orally every 30 minutes, 4 times on the day of surgery.
  Starting from the first day after surgery, patients consumed 200 ml of fat-free nutritional liquid (50 g enzymatically hydrolyzed rice powder + 7.5 g isolated whey protein + 0.5 g low-sodium salt; 223 kcal) per serving, 4 to 6 times per day as needed.
  Arms: experimental group

SUMMARY:
Exploring the effects of whey protein combined with carbohydrates in an Enhanced Recovery After Surgery (ERAS) protocol on the postoperative recovery of thyroid cancer patients undergoing lateral neck dissection, aiming to provide more precise research and guidance for the perioperative accelerated recovery plan in such patients. The goal is to accelerate postoperative recovery and reduce postoperative complications for thyroid cancer patients undergoing neck dissection.

DETAILED DESCRIPTION:
Perioperative dietary management was differentiated between the two groups:

Experimental Group:

6 hours before surgery, patients orally consumed 250 ml of a full-nutrition liquid (220 ml homogenized diet, 50 g; containing 31.4 g carbohydrates, 8 g protein, and 215 kcal).

2 hours before surgery, patients orally consumed 200 ml of a clear liquid (50 g enzymatically hydrolyzed rice powder + 0.5 g low-sodium salt; containing 47.7 g carbohydrates, 6.5 g whey protein, and 193 kcal).

After surgery, once there were no symptoms such as dizziness or vomiting, patients could start consuming clear liquids (containing 47.7 g carbohydrates, 6.5 g protein, and 221 kcal) orally every 30 minutes, 4 times on the day of surgery.

Starting from the first day after surgery, patients consumed 200 ml of fat-free nutritional liquid (50 g enzymatically hydrolyzed rice powder + 7.5 g isolated whey protein + 0.5 g low-sodium salt; 223 kcal) per serving, 4 to 6 times per day as needed.

Control Group:

Patients fasted for 12 hours before surgery, and after surgery, intravenous fluids were administered. Fat-free diet began after 24 hours post-surgery.

Discharge Criteria: The discharge time was determined by the surgeon based on the patient's postoperative drainage condition and the presence or absence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Differentiated thyroid cancer with lateral lymph node dissection;
* Written informed consent provided by the participant.

Exclusion Criteria:

* History of chronic liver or kidney disease, ischemic heart disease, or diabetes;
* Previous neck surgery or history of iodine-131 radiation;
* Allergy to soy or whey protein;
* Intraoperative chylous leak;
* Other special types of thyroid cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
hemoglobin | 3 day
  Record the difference in indicators before and after surgery
serum albumin | 3 day
  the difference in indicators before and after surgery.
Postoperative Complication | 1 month
  Record the occurrence of related surgical complications in the experimental group and the control group.
weight | 1week
  Record the difference in indicators before and after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing General Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No